CLINICAL TRIAL: NCT03609892
Title: Rescue Therapy for Helicobacter Pylori Eradication: A Randomized and Non-inferiority Trail of Berberine Plus Amoxicillin Quadruple Therapy Versus Tetracycline Plus Furazolidone Quadruple Therapy
Brief Title: Helicobacter Rescue Therapy With Berberine Plus Amoxicillin Quadruple Therapy Versus Tetracycline Plus Furazolidone Quadruple Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Responsible Party: Principal Investigator, Yongquan Shi, Professor, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20182043-1
Record Dates: First submitted 2018-07-25; First posted 2018-08-01 (Actual); Last update posted 2019-08-30 (Actual); Status verified 2018-07

CONDITIONS: Gastric Ulcer; Chronic Gastritis; Gastric Cancer; Helicobacter Pylori Infection; Gastritis
MeSH Terms: conditions — Stomach Ulcer; Stomach Neoplasms; Gastritis | interventions — Berberine; Amoxicillin; Esomeprazole; Bismuth; Tetracycline; Furazolidone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- berberine plus amoxicillin quadruple therapy (Experimental): Berberine 500mg three time daily for 14days, amoxicillin 1000 mg, esomeprazole 20 mg, and Bismuth 200mg by mouth, twice daily for 14 days.
  Interventions: Drug: Berberine; Drug: Amoxicillin; Drug: Esomeprazole; Drug: Bismuth
- tetracycline plus furazolidone quadruple therapy (Active Comparator): Tetracycline 500mg three time daily for 14days，furazolidone 100 mg, esomeprazole 20 mg, and Bismuth 200mg by mouth, twice daily for 14 days.
  Interventions: Drug: Tetracycline; Drug: Furazolidone; Drug: Esomeprazole; Drug: Bismuth

INTERVENTIONS:
Drug: Berberine — Berberine-amoxicillin quadruple therapy group: given for 14 days at a dose of berberine 100 mg 3 tablets TID, amoxicillin 500 mg 2 capsules BID ，esomeprazole 20 mg BID, ,and Bismuth 100 mg 2 capsules BID.
  Arms: berberine plus amoxicillin quadruple therapy
Drug: Amoxicillin — Berberine-amoxicillin quadruple therapy group: given for 14 days at a dose of Amoxicillin 500 mg 2 capsules BID plus berberine 100 mg 3 tablets TID, esomeprazole 20mg 1tablet BID, and bismuth 100 mg 2 capsules BID
  Other Names: Amoxy
  Arms: berberine plus amoxicillin quadruple therapy
Drug: Esomeprazole — Berberine-amoxicillin quadruple therapy group: given for 14 days at a dose of Esomeprazole 20mg 1 tablet BID plus berberine 100 mg 3 tablets TID,amoxicillin 500 mg 2 capsules BID, and bismuth 100 mg 2 capsules BID
  Other Names: Nexium
  Arms: berberine plus amoxicillin quadruple therapy
Drug: Bismuth — Tetracycline-furazolidone containing quadruple therapy group: given for 14 days at a dose of Tetracycline 250mg 2 capsules TID plus furazolidone 100mg 1 tablets BID，esomeprazole 20 mg 1 tablets BID and bismuth 100 mg 2 capsules BID
  Arms: berberine plus amoxicillin quadruple therapy
Drug: Tetracycline — Tetracycline-furazolidone containing quadruple therapy group: given for 14 days at a dose of Tetracycline 250mg 2 capsulesTID plus furazolidone 100mg 1 tablets BID，esomeprazole 20 mg 1 tablets BID and bismuth 100 mg 2 capsules BID
  Arms: tetracycline plus furazolidone quadruple therapy
Drug: Furazolidone — Tetracycline-furazolidone containing quadruple therapy group: given for 14 days at a dose of furazolidone 100mg 1 tablets BID plus Tetracycline 250mg 2 capsulesTID，esomeprazole 20 mg 1 tablets BID and bismuth 100 mg 2 capsules BID
  Arms: tetracycline plus furazolidone quadruple therapy
Drug: Esomeprazole — Tetracycline-furazolidone containing quadruple therapy group: given for 14 days at a dose of esomeprazole 20 mg 1 tablets BID plus Tetracycline 250mg 2 capsules TID, furazolidone 100mg 1 tablets BID， and bismuth 100 mg 2 capsules BID
  Other Names: Nexium
  Arms: tetracycline plus furazolidone quadruple therapy
Drug: Bismuth — Tetracycline-furazolidone containing quadruple therapy group: given for 14 days at a dose of bismuth 100 mg 2 capsules BID plus Tetracycline 250mg 2 capsules TID ，furazolidone 100mg 1 tablets BID and esomeprazole 20 mg 1 tablets BID
  Arms: tetracycline plus furazolidone quadruple therapy

SUMMARY:
This study aims at evaluating efficacy and safety of berberine- amoxicillin containing quadruple therapy(berberine, amoxicillin, esomeprazole and bismuth) versus tetracycline-furazolidone quadruple therapy (tetracycline, furazolidone, esomeprazole and bismuth) in H. pylori rescue therapy. It is hypothesized that berberine-amoxicillin containing quadruple therapy is non-inferior to tetracycline-furazolidone quadruple therapy. Patients with confirmed failure of H. pylori eradication will be randomized to one of the treatments described above. At week 6 follow-up visits, a urea breath test，rapid urease test or helicobacter pylori stool antigen test will be performed to confirm eradication.

DETAILED DESCRIPTION:
Detailed Description:

The study will include three phases: screening, treatment and follow-up. Screening: this phase will last a maximum of 14 days and subjects eligibility will be evaluated after signing informed consent. One of urea breath test，rapid urease test or helicobacter pylori stool antigen test will be performed in addition to the baseline routine evaluations.

Treatment: Subjects are randomly assigned to treatment and will be treated for 14 days. A randomization visit will take place on Day 0 and an end-of-treatment visit will take place between day 13 and 17.

Follow-up: includes one visits. Approximately 28 days after the end of treatment. Eradication of H. Pylori will be confirmed by one of urea breath test，rapid urease test or helicobacter pylori stool antigen test。

ELIGIBILITY:
Inclusion Criteria:

1. Patients who had failed H.pylori eradication therapies before.
2. Age between 18~70, both gender.
3. Patients who had failed H.pylori eradication therapies during last 2 years and stop the eradication therapies for at least 2 months.
4. Women are eligible if they are not pregnant or nursing, and if they are of childbearing potential they are required to use medically acceptable contraception for the duration of the study and 30 days thereafter.

Exclusion Criteria:

1. Patients are excluded if they have previously used tetracycline and furazolidone antibiotics to eradicate infection with H. pylori.
2. Contraindications to study drugs.
3. Substantial organ impairment, severe or unstable cardiopulmonary or endocrine disease.
4. Constant use of anti-ulcer drugs ( including taking proton-pump. inhibitors(PPI) within 2 weeks before the [13C] urea breath test), antibiotics or bismuth complexes (more than 3 times /1 month before screening).
5. Pregnant or lactating women.
6. Underwent upper gastrointestinal Surgery.
7. Patients with Barrett esophageal or highly atypical hyperplasia, have symptom of dysphagia.
8. Evidence of bleeding or iron efficiency anemia.
9. A history of malignancy.
10. Drug or alcohol abuse history in the past 1 year.
11. Systemic use of corticosteroids, non steroidal anti-inflammatory drugs, anticoagulants, platelet aggregation inhibitors (except the use of aspirin for less than 100 mg/d).
12. Enrolled in other clinical trials in the past 3 months.
13. Patients who has psychological problem or poor compliance.
14. Refuse to sign informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 658 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
Helicobacter pylori eradication | 28 days after treatment
  The primary end point of this study is H.pylori eradication,established by negative urea breath test，rapid urease test or helicobacter pylori stool antigen test 28 days after the end of treatment.

SECONDARY OUTCOMES:
symptoms effective rates | 14 days of treatment, and 28 days after treatment
  Evaluation effective rate of symptoms 2 weeks of treatment and 4 weeks after the end of treatment.
  Symptom effective rate =（total score before treatment - total score after treatment）/total score before treatment x 100%.
  Total score = frequency * severity.
  Frequency score is calculated by all the frequency of heartburn, reflux, abdominal pain, and flatulence.
  Severity is accumulated by the degree of symptoms described above, which is divided to 4 degree as 0 presenting none, and 3 presenting most severe
adverse events | 14 days of treatment, and 28 days after treatment
  Participants with Adverse Events as a Measure of Safety and Tolerability.The common side effects of the study include headache, dizziness, skin rash, other gastrointestinal disorders, pyrexia, cough and back pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hosipital of Digestive Disease, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang J, Han C, Lu WQ, Wang N, Wu SR, Wang YX, Ma JP, Wang JH, Hao C, Yuan DH, Liu N, Shi YQ. A randomized, multicenter and noninferiority study of amoxicillin plus berberine vs tetracycline plus furazolidone in quadruple therapy for Helicobacter pylori rescue treatment. J Dig Dis. 2020 May;21(5):256-263. doi: 10.1111/1751-2980.12870. Epub 2020 Jun 9. PMID 32348007